CLINICAL TRIAL: NCT00534417
Title: Phase II Trial of Capecitabine in Combination With Fulvestrant for Postmenopausal Women With Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Phase II Trial of Capecitabine With Fulvestrant for Postmenopausal Women With Hormone Receptor Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Hoffmann-La Roche (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSSMBC0606
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Hormone; Receptor; Positive; Metastatic; Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Capecitabine; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine and fulvestrant (Experimental): Capecitabine will be given on a continuous basis at a total dose of 1500 mg, given as 1000 mg po AM and 500 mg po PM in patients of body weight < 80 kg, and at a total dose of 2000 mg given as 1000 mg po bid in patients with a body weight of ≥80 kg.
  Fulvestrant will be given at 500 mg on Day 1 followed by 250 mg on Days 15 and 29, then 250 mg every 28 days.
  Interventions: Drug: capecitabine; Drug: fulvestrant

INTERVENTIONS:
Drug: capecitabine — Capecitabine will be given on a continuous basis at a total dose of 1500 mg, given as 1000 mg po in the morning (AM) and 500 mg po in the evening (PM) in patients of body weight < 80 Kg, and at a total dose of 2000 mg given as 1000 mg po bid in patients with a body weight of ≥80 Kg.
  Other Names: Xeloda
Drug: fulvestrant — Fulvestrant will be given at 500mg on Day 1 followed by 250 mg on Days 15 and 29, then 250mg every 28 days(Q28d).
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to determine if the combination of continuous daily capecitabine with fulvestrant on a loading dose schedule will delay disease progression in metastatic breast cancer (MBC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* At least 18 years of age.
* Post-menopausal female (ie, amenorrheic for at least 12 months prior to study entry). Post-menopausal status will be confirmed by drawing follicle stimulating hormone (FSH) and estradiol levels if < 2 years since last menses.
* Ambulatory outpatient with Eastern Cooperative Oncology Group (ECOG)performance status of 0 to 2 at study entry.
* Primary tumor human epidermal growth factor receptor 2 (HER-2) negative at study entry.(Investigator discretion will be used in instances of immuno-histochemistry [IHC] 2+.)
* Histologically or cytologically confirmed MBC.
* Primary tumor and/or metastatic lesion estrogen receptor + and/or progesterone receptor + by IHC.
* At least one measurable or evaluable(non-measurable) lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria (see Appendix 11.6) which has not been irradiated (i.e., newly arising lesions in previously irradiated areas are accepted). Ascites, pleural effusion, and bone metastases are not considered measurable but are considered evaluable (non-measurable). Minimum indicator lesion size for measurable disease: ≥10 mm measured by spiral computed tomography (CT) or ≥20 mm measured by conventional techniques.
* Adequate hematologic, renal, and hepatic function.

  * Hematologic values: Neutrophils (ANC) > 1.5 x 109/L; Platelet count > 100 x 109/L.
  * Renal function: estimated creatinine clearance > 30 mL/min as calculated with Cockcroft-Gault equation.
  * Note: In patients with moderate renal impairment (calculated creatinine clearance 30 to 50 mL/min) at baseline, a dose reduction to (-1) of the capecitabine starting dose is required.
  * Serum bilirubin < 1.5 x upper limit normal (ULN).
  * Alanine transaminase (ALT) or aspartate transaminase (AST) < 2.5 x ULN (or < 5 x ULN in the case of liver metastases).
  * Alkaline phosphatase < 2.5 x ULN (or < 5 x ULN in the case of liver metastases or < 10 x ULN in the case of bone disease).
  * International normalization ratio (INR) < 1.6.
* Must have ≤ 1 prior regimen of endocrine therapy for metastatic breast cancer. This would include patients who have a recurrence while on adjuvant hormone therapy OR have first recurrence after adjuvant hormone therapy OR progressed after first line hormone therapy for metastatic breast cancer OR treatment naïve patients who present with metastatic breast cancer.

Exclusion Criteria:

* Prior administration of capecitabine.
* Prior administration of fulvestrant.
* Prior chemotherapy for metastatic breast cancer.
* Radiotherapy ≤ 2 weeks prior to registration, except if to a non-target lesion only or single-dose radiation for palliation. NOTE: Prior radiation to a target lesion(s) is permitted only if there has been clear progression of the lesion since radiation was completed.
* Life expectancy <3 months.
* Serious, uncontrolled, concurrent infection(s).
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil or known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Treatment for other carcinomas within the last 5 years, except cured non-melanoma skin and treated in-situ cervical cancer or superficial bladder tumors (stage Ta or Tis).
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Clinically significant cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication)or myocardial infarction within the last 12 months prior to study entry.
* Active brain metastases. Patients with neurological symptoms must undergo a CT scan or magnetic resonance imaging (MRI) of the brain to exclude active brain metastasis. NOTE: Patients with treated brain metastases are eligible provided they have no evidence of disease and are off definitive therapy (including steroids) ≥ 3 months prior to study entry.
* Central nervous system (CNS) disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake.
* Known human immunodeficiency virus or chronic hepatitis B or C.
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Lack of physical integrity of the upper GI tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy.
* Any of the following laboratory values:
* Abnormal hematologic values (neutrophils [ANC]: <1.5 × 109/L, platelet count: <100 × 109/L)
* Impaired renal function (estimated creatinine clearance: <30 mL/min as calculated with Cockcroft-Gault equation). Note: In patients with moderate renal impairment (calculated creatinine clearance: 30 to 50 mL/min) at baseline, a dose reduction to (-1) of the capecitabine starting dose is required.
* Serum bilirubin >1.5 × upper normal limit (ULN).
* Alanine transaminase (ALT) or aspartate transaminase (AST) >2.5 × ULN (or >5 × ULN in the case of liver metastases).
* Alkaline phosphatase > 2.5 × ULN (or >5 × ULN in the case of liver metastases or >10 × ULN in the case of bone disease).
* International normalization ratio (INR) >1.6.
* History of:

  * Bleeding diathesis,(ie, disseminated intravascular coagulation [DIC], clotting factor deficiency) or
  * Long-term anticoagulant therapy,(other than antiplatelet therapy and warfarin 1 mg qd for port prophylaxis).
* History of hypersensitivity to active or inactive excipients of fulvestrant (ie, castor oil or Mannitol).
* Unwillingness to give written informed consent.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Schwartzberg, MD, Principal Investigator — Acorn Cardiovascular, Inc.
Locations (10):
- United States (10):
  - Advanced Medical Specialties, Miami, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Augusta Oncology Associates, Augusta, Georgia
  - Medical & Surgical Specialists, Galesburg, Illinois
  - Oncology Specialists, Park Ridge, Illinois
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Las Vegas Cancer Center, Henderson, Nevada
  - The Lancaster Cancer Center, Ltd, Lancaster, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of Tidewater, Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 community oncology research sites across the US associated with ACORN participated in this study. Enrollment started in February 2008 and was completed in May 2010.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent screening procedures to verify eligibility.
Groups:
- Capecitabine and Fulvestrant: Capecitabine will be given on a continuous basis at a total dose of 1500 mg, given as 1000 mg orally (po) in the morning (AM) and 500 mg po in the evening (PM) in patients of body weight < 80 kg, and at a total dose of 2000 mg given as 1000 mg po bid in patients with a body weight of ≥80 kg.
  Fulvestrant will be given at 500 mg on Day 1 followed by 250 mg on Days 15 and 29, then 250 mg every 28 days.
Period: Overall Study
Arm/Group | Capecitabine and Fulvestrant
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Capecitabine/Fulvestrant: Capecitabine will be given on a continuous basis at a total dose of 1500 mg, given as 1000 mg po AM and 500 mg po PM in patients of body weight < 80 kg, and at a total dose of 2000 mg given as 1000 mg po bid in patients with a body weight of ≥80 kg.
  Fulvestrant will be given at 500 mg on Day 1 followed by 250 mg on Days 15 and 29, then 250 mg every 28 days.
Arm/Group | Treatment Group: Capecitabine/Fulvestrant
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from treatment start until objective tumor progression. Progression is defined per Response Evaluation Criteria in Solid Tumors (RECIST)v1.0 guidelines as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions. The median time to progression is the parameter used to describe TTP.
Time Frame: TTP was measured from day 1 of treatment until time of progression (assessed every 8 weeks), up to 29 months.
Population: 21 patients had experienced disease progression. 20 patients were censored in TTP analysis. The 3 deaths in the PFS analysis were censored for the TTP analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 41
Months | 26.94 (1.84) [7.26 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Secondary Outcome: Best Overall Response
Description: Best overall response is defined as the best response across all time points. Response was evaluated via changes from baseline in radiological tumor measurements performed after every two treatment cycles and at the end of treatment or time of progression. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: Response to treatment was assessed after every 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 41
participants
  Complete response (CR) | 2
  Partial response (PR) | 8
  Stable disease (SD) | 28
  Progressive disease (PD) | 3

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants experiencing complete response (CR) and partial response (PR). Response was evaluated via changes from baseline in radiological tumor measurements performed after every two treatment cycles and at the end of treatment or time of progression. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: Response to treatment was assessed after every 8 weeks of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 41
percentage of participants | 24.4 [10.0 to 38.8]

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of participants experiencing stable disease (SD) of at least 24 weeks plus complete response (CR) and partial response (PR). Response was evaluated via changes from baseline in radiological tumor measurements performed after every two treatment cycles and at the end of treatment or time of progression. Response was evaluated using RECIST version 1.0 guidelines, where CR is the disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter(LD) of target lesions; SD is neither sufficient shrinkage in sum of longest diameter of target lesions to be PR nor increase of >=20%.
Time Frame: Response to treatment was assessed after every 8 weeks of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 41
percentage of participants | 58.5 [42.2 to 73.3]

5. Primary Outcome: Progression-free Survival (PFS)
Description: Disease progression was determined through radiology imaging measurements and by clinical or symptomatic progression during or after treatment. Progression is defined per RECIST v1.0 guidelines as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: PFS was measured from day 1 of treatment until time of progression (assessed every 8 weeks) or death, whichever came first, up to 32.5 months.
Population: 21 patients had experienced disease progression, and three had died. 17 patients were censored in PFS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 41
Months | 14.98 [7.26 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

6. Secondary Outcome: Patients Experiencing Severe Symptom Burden (Physical Symptoms)
Description: The subject rates each question about physical symptoms on a scale of 0 through 10, where 0 is not bad and 10 is as bad as possible. Severe symptoms are indicated by a response > or = to 7 on an item.
Time Frame: The questionnaire was administered on day 1 of every cycle (approximately every 4 weeks) during study treatment.
Population: Participants who had questionnaire data available.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 30
percentage of participants
  Hives/Welts | 3.3
  Sinus problems | 3.3
  Swelling | 10.0
  Fatigue | 26.7
  Weight loss | 10.0
  Change in taste | 6.7
  Difficulty hearing | 3.3
  Reduced sexual enjoyment, interest, or performance | 10.0
  Dry eyes | 10.0
  Tearing | 10.0
  Trouble seeing | 16.7
  Constipation | 20.0
  Decrease in appetite | 6.7
  Diarrhea | 3.3
  Heartburn | 6.7
  Increase in appetite | 3.3
  Problem with urination | 3.3
  Vaginal dryness | 3.3
  Bruising | 3.3
  New lump/mass | 6.7
  Breast tenderness | 3.3
  Dry skin | 13.3
  Hair loss | 3.3
  Itching | 13.3
  Nails change | 10.0
  Joint pain | 26.7
  Muscle aches | 26.7
  Weakness of body parts | 10.0
  Burning sensation in hands or feet | 10.0
  Daytime sleepiness | 10.0
  Dizziness/lightheadedness | 3.3
  Memory loss | 6.7
  Numbness/tingling | 13.3
  Trouble thinking | 10.0
  Headache | 6.7
  Pain | 26.7
  Coughing | 13.3
  Shortness of breath | 6.7
  Wheezing | 6.7

7. Secondary Outcome: Patients Experiencing Severe Symptom Burden (Psychiatric Symptoms)
Description: The subject rates each question about psychiatric symptoms on a scale of 0 through 10, where 0 is not bad and 10 is as bad as possible. Severe symptoms are indicated by a response > or = to 7 on an item.
Time Frame: The questionnaire was administered on day 1 of every cycle (approximately every 4 weeks) during study treatment.
Population: Participants who had questionnaire data available.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 29
percentage of participants
  Crying/feeling like crying | 10.3
  Feeling helpless | 6.9
  Feeling hopeless | 10.3
  Feeling I would be better off dead | 3.4
  Lost interest in people | 3.4
  Lost interest in pleasurable activities | 10.3
  Nervous, tense, anxious | 13.8
  Sad/depressed | 10.3
  Worry | 10.3

8. Post Hoc Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death from any cause. The median overall survival time is used to measure OS.
Time Frame: OS was measured from day 1 of treatment until time of death from any cause, up to 32.5 months.
Population: 14 patients had died, and 27 patients were censored in the OS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 41
Months | 28.65 [23.95 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

9. Secondary Outcome: Patients Experiencing Severe Symptom Burden (Physical Functioning)
Description: The subject rates each question about physical functioning on a scale of 0 through 10, where 0 is not bad and 10 is as bad as possible. Severe symptoms are indicated by a response > or = to 7 on an item.
Time Frame: The questionnaire was administered on day 1 of every cycle (approximately every 4 weeks) during study treatment.
Population: Participants who had questionnaire data available. Note that 4 items only had data available from 27 participants rather than 28.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine and Fulvestrant
Number analyzed (Participants) | 28
percentage of participants
  Attend paid job (N=27) | 37.0
  Attend social activity | 7.1
  Bathe or dress self | 10.7
  Cook for self | 10.7
  Driving (N=27) | 25.9
  Function normally | 14.3
  Hard work or activity (N=27) | 33.3
  Household work | 21.4
  Light work or activity | 10.7
  Run (N=27) | 33.3
  Run errands | 17.9
  Sit up | 10.7
  Stay out of bed | 7.1
  Walk | 17.9

ADVERSE EVENTS:
Time Frame: Adverse events were collected on day 1 of treatment until one month after the end of study treatment.
Arm/Group | Treatment Group: Capecitabine/Fulvestrant
Serious Adverse Events (participants affected / at risk) | 9/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: Capecitabine/Fulvestrant (N=41)
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac Tamponade (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Adverse Drug Reaction (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Hepatic Enzyme Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Cerebrovascular Accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group: Capecitabine/Fulvestrant (N=41)
Anaemia (Blood and lymphatic system disorders) | 4
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Cerumen Impaction (Ear and labyrinth disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Diplopia (Eye disorders) | 2
Dry Eye (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Lacrimation Increased (Eye disorders) | 3
Vision Blurred (Eye disorders) | 1
Visual Impairment (Eye disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 10
Dry Mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Rectal Haemorrhage (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 4
Axillary Pain (General disorders) | 2
Chest Discomfort (General disorders) | 2
Chest Pain (Gastrointestinal disorders) | 4
Chills (General disorders) | 2
Device Occlusion (General disorders) | 1
Face Oedema (General disorders) | 1
Fatigue (General disorders) | 16
Gait Disturbance (General disorders) | 1
Immediate Post-Injection Reaction (General disorders) | 2
Influenza Like Illness (General disorders) | 1
Injection Site Pain (General disorders) | 1
Injection Site Pruritus (General disorders) | 2
Mucosal Inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 10
Pain (General disorders) | 3
Pyrexia (General disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Fungal Skin Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 5
Vaginal Infection (Infections and infestations) | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Joint Injury (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Decreased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 3
Blood Pressure Increased (Investigations) | 1
Breath Sounds Abnormal (Investigations) | 1
Creatinine Renal Clearance Increased (Investigations) | 1
Heart Rate Increased (Investigations) | 1
Protein Total Decreased (Investigations) | 1
Prothrombin Level Increased (Investigations) | 1
Prothrombin Time Prolonged (Investigations) | 1
Thyroid Function Test Abnormal (Investigations) | 1
Vitamin D Decreased (Investigations) | 1
Weight Decreased (Investigations) | 2
Weight Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7
Increased Appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck Mass (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 9
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Burning Feet Syndrome (Nervous system disorders) | 1
Burning Sensation (Nervous system disorders) | 2
Cerebral Ischaemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 2
Mental Impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Restless Legs Syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sinus Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 3
Urinary Retention (Renal and urinary disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 2
Vaginal Haemorrhage (Reproductive system and breast disorders) | 2
Vulvovaginal Dryness (Reproductive system and breast disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Discharge Discolouration (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 3
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1
Increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 2
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 8
Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Skin Mass (Skin and subcutaneous tissue disorders) | 1
Skin Sensitisation (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4
Deep Vein Thrombosis (Vascular disorders) | 2
Hot Flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall submit a copy of any manuscript or material proposed for publication or the text of any presentation relating to the results of the Study to AstraZeneca and Roche for review and comment at least 30 days prior to its submission for publication or presentation.